CLINICAL TRIAL: NCT02338765
Title: With Help From Buddies: The Impact of Social Support Using Mobile Technology on Physical Activity Among Women With Young Children
Brief Title: MoTHER Buddy Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, JiWon Choi, Assistant Adjunct Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A123858
Record Dates: First submitted 2015-01-07; First posted 2015-01-14 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Physical Activity; Obesity
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buddy (Experimental): Physical activity plus having a buddy
  Interventions: Behavioral: mHealth Physical Activity; Behavioral: Buddy-partnered exercise
- Control (Active Comparator): Physical activity only
  Interventions: Behavioral: mHealth Physical Activity

INTERVENTIONS:
Behavioral: mHealth Physical Activity
Behavioral: Buddy-partnered exercise
  Arms: Buddy

SUMMARY:
The purpose of the 12-week study is to determine if competing a physical activity program with a buddy helps increase daily physical activity when compared to completing the same physical activity program without a buddy.

ELIGIBILITY:
Inclusion Criteria:

1. Physically inactive,
2. having at least one child aged less than 5 years,
3. having at least one family member or friend who can support physical activity engagement and reside in the same community,
4. having access to computer and phone, and
5. overweight/obese (Body Mass Index: 23 kg/m2 or more)

Exclusion Criteria:

1. Having known medical conditions that prevent regular physical activity and
2. current participation in other lifestyle modification programs

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Daily steps | weekly during study period, up to 12 weeks

SECONDARY OUTCOMES:
Weight | Changes in weight over the 12-week study period
Waist Circumference (WC) | Changes in WC over the 12-week study period
Hip Circumference (HC) | Changes in HC over the 12-week study period

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States